CLINICAL TRIAL: NCT02908230
Title: Camp NERF: Methods of a Theory-Based Nutrition Education Recreation and Fitness Program Aimed at Preventing Unhealthy Weight Gain in Underserved Elementary Children During Summer Months
Brief Title: Camp NERF: Methods of a Summer Nutrition Ed Rec & Fitness Program to Prevent Unhealthy Weight Gain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Aetna Foundation (Unknown)
Responsible Party: Principal Investigator, Carolyn Gunther, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014B0197
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Control (Placebo Comparator): Active Control: exposure to a non-nutrition, physical activity, or mental health curriculum/program
  Interventions: Behavioral: Active Control
- Standard Care (Active Comparator): Standard Care: exposure to a nutrition and physical activity curriculum/program
  Interventions: Behavioral: Standard Care
- Enhanced Care (Experimental): Enhanced Care: exposure to a nutrition, physical activity, and mental health curriculum/program
  Interventions: Behavioral: Enhanced Care

INTERVENTIONS:
Behavioral: Enhanced Care — 8-week (nutrition, physical activity, and mental health) summer curriculum/program
  Arms: Enhanced Care
Behavioral: Standard Care — 8-week (nutrition and physical activity) summer curriculum/program
  Arms: Standard Care
Behavioral: Active Control — 8-week (non-nutrition, physical activity or mental health) summer curriculum/program
  Arms: Active Control

SUMMARY:
The primary aims of this research project are to:

1. Evaluate the efficacy of Camp NERF to improve child nutrition, physical activity, mental health, and anthropometric outcomes.
2. Evaluate the efficacy of Camp NERF to improve caregiver self-efficacy for establishing healthy family nutrition and physical activity practices, amount of physical activity, and BMI.
3. Evaluate the efficacy of Camp NERF to improve youth mentor nutrition, physical activity, and anthropometric outcomes.

DETAILED DESCRIPTION:
Background: The number of obese children in the US remains high, which is problematic due to the mental, physical, and academic effects of obesity on child health. Data indicate that school-age children, particularly underserved children, experience unhealthy gains in BMI at a rate nearly twice as fast during the summer months. Few efforts have been directed at implementing evidence-based programming to prevent excess weight gain during the summer recess.

Methods: Camp NERF is an 8-week, multi-component (nutrition, physical activity, and mental health), theory-based program for underserved school-age children in grades Kindergarten - 5th grade coupled with the USDA Summer Food Service Program. Twelve eligible elementary school sites will be randomized to one of the three programming groups: 1) Active Control (non-nutrition, physical activity, or mental health [4H curricula]); 2) Standard Care (nutrition and physical activity); or 3) Enhanced Care (nutrition, physical activity, and mental health) programming. Anthropometric, behavioral, and psychosocial data will be collected from child-caregiver dyads pre- and post-intervention. Site-specific characteristics and process evaluation measures will also be collected.

Discussion: This is the first, evidence-based intervention to address the issue of weight gain during the summer months among underserved, school-aged children. Results from this study will provide researchers, practitioners, and public health professionals with insight on evidence-based programming to aid in childhood obesity prevention during this particular window of risk.

ELIGIBILITY:
Inclusion Criteria (site level):

* Elementary school; USDA Summer Food Service Program open site; and 3) lacking structured programming

Exclusion Criteria:

-

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in child BMI z-score | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn W Gunther, PhD, Principal Investigator — Ohio State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hopkins LC, Webster A, Kennel JA, Purtell KM, Gunther C. Youth Mentor Dietary Outcomes and Waist Circumference Improvement: Camp NERF Study Findings. Health Promot Pract. 2020 Nov;21(6):962-971. doi: 10.1177/1524839919833989. Epub 2019 Feb 28. PMID 30819010
- [Derived] Hopkins LC, Fristad M, Goodway JD, Melnyk B, Eneli I, Holloman C, Kennel JA, Webster A, Sharn AR, Gunther C. Feasibility and acceptability of technology-based caregiver engagement strategies delivered in a summertime childhood obesity prevention intervention: results from an internal pilot of the Camp NERF (Nutrition, Education, Recreation, and Fitness) study. Pilot Feasibility Stud. 2018 Sep 27;4:153. doi: 10.1186/s40814-018-0340-2. eCollection 2018. PMID 30275966
- [Derived] Hopkins LC, Fristad M, Goodway JD, Eneli I, Holloman C, Kennel JA, Melnyk B, Gunther C. Camp NERF: methods of a theory-based nutrition education recreation and fitness program aimed at preventing unhealthy weight gain in underserved elementary children during summer months. BMC Public Health. 2016 Oct 26;16(1):1122. doi: 10.1186/s12889-016-3765-7. PMID 27784290